CLINICAL TRIAL: NCT05789888
Title: Evaluation of the Influence of SNP Variability of Stearoyl-CoA Desaturase (SCD) Gene of Nuclear DNA and MT-ATP6 Gene of Mitochondrial DNA and Environmental Factors on Phenotypic Variability of Visceral and Subcutaneous Adipose Tissue
Brief Title: Genes Variability in Obesity and Normal Body Weight Patients.
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: SUB/3/DN/22/001/3316
Record Dates: First submitted 2023-03-08; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Obesity, Visceral; Obesity
Keywords: SCD; MT-ATP6; Obesity; VAT; SAT; TOFI; FOTI; Genetic; Genes; Phenotype
MeSH Terms: conditions — Obesity, Abdominal; Obesity | interventions — Adiposity; Phenotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Swabs from mouth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: The study group consisted of 75 people (46 women and 29 men) with gender (BMI=30.0-39.9 kg/m2).
  Interventions: Genetic: MT-ATP6 mtDNA gene variability in obesity and normal body weight patients.; Genetic: SCD gene variability in obesity and normal body weight patients.; Other: Finding TOFI and FOTI phenotypes in participants with obesity and normal weight.
- Control group: The control group included 41 people (31 women and 10 men) with normal weight (BMI=18.5-24.9 kg/m2).
  Interventions: Genetic: MT-ATP6 mtDNA gene variability in obesity and normal body weight patients.; Genetic: SCD gene variability in obesity and normal body weight patients.; Other: Finding TOFI and FOTI phenotypes in participants with obesity and normal weight.

INTERVENTIONS:
Genetic: MT-ATP6 mtDNA gene variability in obesity and normal body weight patients. — As part of the research, the MT-ATP6 gene was tested in order to influence the modulation of the amount of fat contained.
  Other Names: The search for obesity markers
Genetic: SCD gene variability in obesity and normal body weight patients. — As part of the research, the SCD gene was tested in order to influence the modulation of the amount of fat contained.
  Other Names: The search for obesity markers
Other: Finding TOFI and FOTI phenotypes in participants with obesity and normal weight. — As part of the research, we measured the amount of VAT and SAT and calculate VAT/SAT ratio as a marker to determine the phenotype of fat tissue.
  Other Names: Phenotypes in obesity

SUMMARY:
The goal of this clinical trial is to learn about variability of gene SCD and MT-ATP6 in describe participant population and health conditions. The main questions it aims to answer are:

• whether there is variation in genes between obese and normal weight individuals

Participants will get body weight and high was assessed using the medical scale and stadiometer, then, basis on obtained results, the Body Mass Index (BMI) will be calculated. Next, participants get determine the body composition and body composition analysis by bioelectrical impedance method to determined: Visceral Adipose Tissue (VAT in cm2 and %), Subcutaneous Adipose Tissue (SAT in cm2 and %), and the VAT/SAT ratio was also determined. Then order to examine the sequence of the genes, swab will take from the oral cavity (cheeks and palate) using sterile swab. The research was carried out at the Department of Dietetics and Clinical Nutrition (Medical University of Bialystok).

DETAILED DESCRIPTION:
The approved of the Bioethics Committee of the Medical University, No. APK.002.407.2020, was obtained for the study. 116 people meeting the inclusion criteria were included in the intervention and observational study. The research was carried out at the Department of Dietetics and Clinical Nutrition at the Faculty of Health Sciences of the Medical University of Bialystok.

The study took place from the April to the September 2021. The analysis were performed in the morning, fasting, without intensive physical ac-tivity. Body weight and high was assessed using the medical scale and stadiometer with an accuracy of 0.01 kg for the body weight and 0.5 cm for the body high. Then, basis on obtained results, the Body Mass Index (BMI) was calculated.Basis on the obtained results the participants were divided into the study group (n=75) and control group (n=41). The study group consisted 46 women and 29 men with primary obesity (BMI=30.0-39.9 kg/m2). The control group consisted 31 women and 10 men with normal body weight (BMI=18.5-24.9 kg/m2).

In order to determine the body composition of participants, a body composition analysis by bioelectrical impedance method was conducted, which enabled the assessment of the following parameters: total body fat mass (kg), total percentage of body fat (%), total percentage of free fat mass (%). The area of adipose tissue in the transverse section to the abdomen was also deter-mined: Visceral Adipose Tissue (VAT in cm2 and %), Subcutaneous Adipose Tissue (SAT in cm2 and %), and the VAT/SAT ratio was also determined. To determine the TOFI phenotype of abdominal fat distribution VAT/SAT ratio was used- above 1 for men and above 0.9 for women.

Next swab from the oral cavity was took. To isolate DNA from the swabs, was used ready kit from A&A Biotechnology. After it we did the PCR reactions with the appropriate primers and clean up after PCR reaction was did. Next we prepared the samples for Sanger sequencing.

When we get the sequences, we used the genetics programs: Bioedit, Chromas, DnaSP, Arlequin, Mega, Genepop to get number of haplotypes, genes variability, F statistics, haplotype diversity, haplotypes network and genetic tree of haplotypes.

ELIGIBILITY:
Inclusion Criteria:

* primary obesity and normal body weight

Exclusion Criteria:

* absence of inflammation and periodontal disease in the oral cavity
* secondary obesity
* type 1 diabetes
* type 2 diabetes
* endocrine disorders
* appetite disorders
* pregnancy and lactation
* acute coronary artery disease
* use of hormonal contraception or hormone replacement therapy
* steroid therapy
* antiretroviral therapy, previous surgical or pharmacological treatment for obesity and pacemaker

Ages: 20 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Inhabitants of the Podlaskie Voivodeship.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
SCD variability between study and control group. | 1 day
  Variability between groups will be determined based on the SCD gene sequence.
MT-ATP6 gene variability. | 1 day
  Variability between groups will be determined based on the MT-ATP6 gene sequence.
Numbers of TOFI and FOTI phenotypes. | 1 day
  On the basis of the VAT/SAT ratio, the abdominal adipose tissue phenotype will assessed.
Genetic variability between TOFI and FOTI phenotypes. | 1 day
  Genetic variability between TOFI and FOTY phenotypes will be determined based on the SCD and MT-ATP6 genes.

CONTACTS AND LOCATIONS:
Overall Officials: Damian D Pogodziński, Master, Study Chair — Medical University of Białystok
Locations (1):
- Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Participants were coded and their IPD will not shared to other reasearchers.